CLINICAL TRIAL: NCT00987714
Title: Monitoring Organ Donors to Increase Transplantation Results
Brief Title: Monitoring Organ Donors to Increase Transplantation Results (MOnIToR)
Acronym: MOnIToR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, John Kellum, M.D., University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R38OT10587
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Transplantation
Keywords: Organ Donors; Recipients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protocolized Care (Experimental): Algorithm to manage Pulse Pressure Variation, Cardiac Index, and Mean Arterial Pressure will be used in these donors.
  Interventions: Procedure: Protocolized care
- Standard Care (No Intervention): This is the Organ Procurement Organization current practices.

INTERVENTIONS:
Procedure: Protocolized care — Organ Procurement Coordinators will utilize a hemodynamic monitor and algorithm for donor management of cardiac index, pulse pressure variation and mean arterial pressure.
  Arms: Protocolized Care

SUMMARY:
The objective of this study is to determine whether protocol guided resuscitation of brain dead organ donors using Pulse Pressure Variation (PPV) will increase the number of organs transplanted per donor.

Specifically the study aims to:

1. improve resuscitation of potential organ donors.
2. improve organ function in donors.
3. increase organ recovery per donor.

The investigators will randomize 960 subjects to either protocolized resuscitation (n=480) using a consensus-based PPV-guided algorithm or usual care using a 1:1 randomization scheme. The primary outcome is the mean number of organs transplanted per donor. Secondary outcomes include 6mHFS (six-month hospital-free survival) in the recipients, and mean number of organs procured per donor that are suitable for transplantation (intention to transplant). The study is powered to detect a 0.5 organ increase for transplantation per donor.

ELIGIBILITY:
Inclusion Criteria:

* Donors who were declared brain dead per local hospital brain death criteria.
* Donors who are deemed suitable for organ donation by the local OPO whether they meet the standard criteria or the extended criteria for donation.
* Presence of functioning arterial catheter.

Exclusion criteria:

* Inability to obtain informed consent from donor next of kin or legal representative.
* Donors less than 16 years of age, no maximum age limit.
* Inability to perform hemodynamic monitoring.
* Patients on lithium therapy prior to brain death.
* Known severe aortic regurgitation, intra-cardiac shunts, or on intra-aortic balloon pump.
* Donors previously enrolled in experimental protocol in which cytokines are the therapeutic targets (e.g. anti-TNF antibodies).
* Donors receiving chemotherapy or with any disease state (e.g. AIDS) that renders the subject leukopenic (WBC count < 2).
* Donors receiving anti-leukocyte drugs (e.g. OKT3) regardless of their WBC counts.
* Pregnant donors.
* Donor is on ECMO machine

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 556 (Actual)
Dates: Start 2009-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Number of organs transplanted. | At explantation

SECONDARY OUTCOMES:
Number of organs that are transplantable. | At Explantation
Expected Observed Ratio | At Explantation
Organ Recipient six month hospital free survival | 6 months post transplant

CONTACTS AND LOCATIONS:
Overall Officials: John Kellum, MD, Principal Investigator — University of Pittsburgh
Locations (8):
- United States (8):
  - LifeLink of Georgia, Norcross, Georgia
  - LifeBanc, Cleveland, Ohio
  - Lifeline of Ohio, Columbus, Ohio
  - LifeShare of Oklahoma, Oklahoma City, Oklahoma
  - Center for Organ Recovey and Education, Pittsburgh, Pennsylvania
  - Tennessee Donor Services, Knoxville, Tennessee
  - Southwest Transplant Alliance-Dallas, Dallas, Texas
  - Lifecenter North West, Bellevue, Washington

REFERENCES:
- [Background] Al-Khafaji A, Murugan R, Wahed AS, Lebovitz DJ, Souter MJ, Kellum JA; MOnIToR study investigators. Monitoring Organ Donors to Improve Transplantation Results (MOnIToR) trial methodology. Crit Care Resusc. 2013 Sep;15(3):234-40. PMID 23944211
- [Result] Al-Khafaji A, Elder M, Lebovitz DJ, Murugan R, Souter M, Stuart S, Wahed AS, Keebler B, Dils D, Mitchell S, Shutterly K, Wilkerson D, Pearse R, Kellum JA. Protocolized fluid therapy in brain-dead donors: the multicenter randomized MOnIToR trial. Intensive Care Med. 2015 Mar;41(3):418-26. doi: 10.1007/s00134-014-3621-0. Epub 2015 Jan 13. PMID 25583616
- [Derived] Li S, Wang S, Murugan R, Al-Khafaji A, Lebovitz DJ, Souter M, Stuart SRN, Kellum JA; Monitoring Organ Donors to Improve Transplantation Results (MOnIToR) Study Investigators. Donor biomarkers as predictors of organ use and recipient survival after neurologically deceased donor organ transplantation. J Crit Care. 2018 Dec;48:42-47. doi: 10.1016/j.jcrc.2018.08.013. Epub 2018 Aug 18. PMID 30172032